CLINICAL TRIAL: NCT00056914
Title: Development of 7 Tesla MRI Methodology for Anatomical Functional and Spectroscopic Imaging of the Brain
Brief Title: Development of Techniques for Use in MRI With a Magnetic Field of 7 Tesla
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030142; 03-N-0142
Record Dates: First submitted 2003-03-26; First posted 2003-03-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-01-05

CONDITIONS: Healthy; Magnetic Resonance Imaging
Keywords: Magnetic Resonance Imaging; Functional Imaging; Cerebral Blood Flow; Parallel Imaging; BOLD Effect; Spectroscopic Imaging; Healthy Volunteer; HV

SUMMARY:
This study will develop new techniques for optimizing resolution in magnetic resonance imaging (MRI) with a high magnetic field of 7 Tesla. MRI is a diagnostic tool that generates high-quality images of the body without the use of x-rays. It can also provide information about brain chemistry and physiology. The test is routinely done at magnetic field strengths of from 1.5 to 4 Tesla. This study will use an investigational device that operates at a high magnetic field of 7 Tesla. Except for the increase in magnetic field, all other aspects of imaging are the same as those at lower magnetic fields. This study will use techniques in conjunction with the higher magnetic field that may improve diagnostic imaging. The MRI will monitor the brain at high resolution to see structural features, to measure brain chemicals, and to determine how much and how fast blood flows into brain regions in response to simple tasks.

Healthy normal volunteers 18 years of age and older may participate in this study. Candidates will be screened with a medical history, neurological examination, and questionnaire.

Participants will have a standard 1.5 or 3 Tesla MRI before the 7 Tesla scan, adding about 5 minutes to the procedure. The procedure for both scans is the same. The subject lies on a table that is moved into the scanner. Because the machine makes loud sounds during the imaging, earplugs are provided to help reduce the noise. An insulated wire coil may be placed around the subject's head to obtain better images. Scanning time varies from 20 minutes to 3 hours, with most examinations lasting between 45 and 90 minutes. During the scan, the subject may be asked to perform simple tasks, such as listening to tones, tapping fingers, moving a hand, watching a movie on a screen, or smelling pleasant odors. More complex tasks may require thinking about tones or pictures and responding to them by pressing buttons. Following the test, subjects will complete a brief questionnaire about comfort level and any unusual sensations they may have experienced during the test.

Participants who undergo repeated MRIs for the evaluation of new techniques will have a standard 1.5 or 3 Tesla MRI brain study once a year while participating in the research protocol. A radiologist at NIH will read the MRIs, and if any abnormalities are discovered, the individual will be referred to his or her private physician or to a consult service at NIH.

...

DETAILED DESCRIPTION:
The goal of this protocol is to optimize new technology that enables Magnetic Resonance Imaging (MRI) at a static magnetic field strength of 7 Tesla (7T). Techniques will be developed for anatomical, functional, and spectroscopic MRI that can take advantage of this high field. Routine clinical MRI has been performed at 1.5T for over twenty years and over the past ten years MRI at 3-4T has demonstrated large increases in sensitivity and is beginning to find widespread application for functional imaging of the brain and clinical research. Since the late 1990's it has been possible to produce magnets with field strengths between 7-9T large enough for human use. Indeed there are presently two sites with 7T and one with 8T MRI that have begun to produce exciting images. These initial results confirm that MRI can be performed safely at these high field strengths and that the whole range of MRI experiments can be performed. We will take delivery of the first 7T MRI system produced by General Electric, the leading producer of MRI equipment, sometime in late 2002/early 2003.

Compared to 3-4T, the 7T scanner is expected to improve sensitivity by a factor of two and improve contrast to noise for functional imaging and spectroscopy by a factor of two - four. However, realizing these goals for routine practice and whole brain coverage will require technical developments and integrating these developments into optimized data acquisition and processing strategies. Therefore, we plan to extend parallel imaging strategies, currently becoming available for 3T MRI, to 7T in order to realize the full gain in sensitivity and apply these techniques to obtain high resolution anatomical MRI, generate high temporal and spatial resolution perfusion images using arterial spin labeling techniques, generate high-temporal and spatial resolution functional images of the brain using blood oxygenation (BOLD) and perfusion based techniques, and test the usefulness of 7T for spectroscopic studies of metabolites of the brain. All of these developments will be performed on normal, healthy volunteers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Only neurologically and psychiatrically normal, male or female, healthy volunteers over 18 years old will be used in these studies. Subjects must be capable of understanding the procedures and requirements of this study. Subjects must be willing to sign an informed consent document.

EXCLUSION CRITERIA:

A subject will be excluded if he/she has a contraindication to MR scanning such as the following: pregnancy, aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or auto-defibrillator; cochlear implant; ocular foreign body (e.g. metal shavings or insulin pump), dental work such as crowns or bridges with indeterminate metals, pre-existing eye conditions, and any pre-existing hearing problems. Subjects who underwent brain surgery, who have a neurological lesion, a psychiatric history or a history of migraine will also be excluded from this study. The contraindications for MRI at 7T are identical to those at 1.5T and 3T.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-03-21; Study Completion 2010-01-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Robitaille PM, Abduljalil AM, Kangarlu A, Zhang X, Yu Y, Burgess R, Bair S, Noa P, Yang L, Zhu H, Palmer B, Jiang Z, Chakeres DM, Spigos D. Human magnetic resonance imaging at 8 T. NMR Biomed. 1998 Oct;11(6):263-5. doi: 10.1002/(sici)1099-1492(199810)11:63.0.co;2-0. PMID 9802467
- [Background] Abduljalil AM, Kangarlu A, Zhang X, Burgess RE, Robitaille PM. Acquisition of human multislice MR images at 8 Tesla. J Comput Assist Tomogr. 1999 May-Jun;23(3):335-40. doi: 10.1097/00004728-199905000-00001. PMID 10348433
- [Background] Burgess RE, Yu Y, Abduljalil AM, Kangarlu A, Robitaille PM. High signal-to-noise FLASH imaging at 8 Tesla. Magn Reson Imaging. 1999 Oct;17(8):1099-103. doi: 10.1016/s0730-725x(99)00072-7. PMID 10499671